CLINICAL TRIAL: NCT04430114
Title: DediCated MuLtibranchEd DacrOn Graft for OPen RepAir of ThoRacoabdominal Aneurysms - CLEOPATRA Study
Brief Title: MuLtibranchEd Graft for OPen RepAir of ThoRacoabdominal Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLEOPATRA study
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aneurysm Abdominal; Aneurysm Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAAA spinal loop graft (Experimental)
  Interventions: Device: branched prosthesis for surgical treatment of thoraco-abdominal aortic aneurysms

INTERVENTIONS:
Device: branched prosthesis for surgical treatment of thoraco-abdominal aortic aneurysms — Jotec "TAAA spinal loop graft" "custom made CE equivalent" branched prosthesis, compared with the cohort of patients already treated with standard prostheses and / or Gelweave ™ Coselli Thoracoabdominal Grafts.

SUMMARY:
The objective of the study is the evaluation of the technical success and clinical outcomes of the surgical treatment of thoraco-abdominal aortic aneurysms treated by Jotec "TAAA spinal loop graft" "custom made "CE equivalent" branched prosthesis, compared with the patient cohort already treated with standard and / or bench-top prostheses Gelweave ™ Coselli Thoracoabdominal Grafts.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years;
* patients candidates for surgical treatment of thoraco-abdominal aorta of the II and III type sec. Crawford using "TAAA spinal loop graft" "custom made CE equivalent" prosthesis

Exclusion Criteria:

• patients aged ≤ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
number of participants who obtain technical success | 12 month
  number of surviving participants
incidence of thrombosis of the prosthetic branches, visceral arteries and replanted intercostal arteries | 12 month
  freedom from thrombosis of the prosthetic branches,visceral arteries and replanted intercostal arteries
incidence of aneurysmal dilatation of visceral and replanted intercostal arteries | 12 month
  freedom from surgical / endovascular reoperation for aneurysmal dilatation of visceral and replanted intercostal arteries

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided